CLINICAL TRIAL: NCT06681649
Title: Improving Medical and Psychological Outcomes After Discharge - Feasibility Study for a Pragmatic, Mixed-methods, Open-label Randomized Controlled Trial Examining the Effectiveness of a Follow-up Clinic for ICU Survivors and Caregivers
Brief Title: Pilot Feasibility Study of a Pragmatic Mixed-Methods Randomized Controlled Trial on a Follow-Up Bundle of Care for ICU Survivors and Caregivers
Acronym: IMPACT-ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Gordon Boyd, Associate Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 6039808
Record Dates: First submitted 2024-10-28; First posted 2024-11-08 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Critical Illness; Delirium in the Intensive Care Unit
Keywords: critical illness; delirium; post-intensive care syndrome
MeSH Terms: conditions — Critical Illness; Delirium; postintensive care syndrome | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive follow-up care through the specialized post-ICU follow-up clinic at KHSC at approximately 1- and 3-months following ICU discharge. Caregivers will also be invited to participate in the follow-up clinic along with the ICU survivor participant.
  In addition to receiving specialized follow-up clinical care, ICU survivor participants and their caregivers will also receive the following additional items as part of a bundled care intervention program (see Appendix):
  * Informational pamphlet on critical illness and expectations following ICU discharge
  * Flyer on critical illness and expectations following ICU discharge (brief version, which may be placed on the participant's refrigerator or other location at home as a consistent reminder)
  * Diaries in which the healthcare team, family members, and the patient themselves are able to journal their experiences, updates, progress, and barriers in the ICU and following discharge
  Interventions: Behavioral: Intervention
- Control (No Intervention): The control group will receive generalized standard of care follow-up through their primary care provider. This follow-up is highly variable depending on the patient and their primary care provider.

INTERVENTIONS:
Behavioral: Intervention — The intervention group will receive follow-up care through the specialized post-ICU follow-up clinic at KHSC at approximately 1- and 3-months following ICU discharge. Caregivers will also be invited to participate in the follow-up clinic along with the ICU survivor participant.
  In addition to receiving specialized follow-up clinical care, ICU survivor participants and their caregivers will also receive the following additional items as part of a bundled care intervention program (see Appendix):
  * Informational pamphlet on critical illness and expectations following ICU discharge
  * Flyer on critical illness and expectations following ICU discharge (brief version, which may be placed on the participant's refrigerator or other location at home as a consistent reminder)
  * Diaries in which the healthcare team, family members, and the patient themselves are able to journal their experiences, updates, progress, and barriers in the ICU and following discharge
  Arms: Intervention

SUMMARY:
~80% of ICU survivors experience profound long-term cognitive, physical, and psychiatric impairments known as post-intensive care syndrome (PICS). Caregivers additionally experience similar detrimental psychosocial effects following discharge. Despite this knowledge, follow-up care is almost non-existent. ICU follow-up clinics may mitigate these long-term impacts, but lack evaluation of their effectiveness. This trial will evaluate the effectiveness of ICU follow-up clinics vs. standard-of-care in improving qualitative/clinical outcomes of ICU survivors and caregivers, with those receiving follow-up care hypothesized to have improved outcomes.

DETAILED DESCRIPTION:
~80% of ICU survivors experience profound long-term cognitive, physical, and psychiatric impairments known as post-intensive care syndrome (PICS), with patients experiencing prolonged delirium or mechanical ventilation having a heightened risk. Caregivers additionally experience similar detrimental psychosocial effects following discharge. Despite this knowledge, follow-up care is almost non-existent. ICU follow-up clinics may mitigate these long-term impacts, but lack evaluation of their effectiveness. This pragmatic, mixed-methods, open-label randomized (1:1) controlled trial will evaluate the effectiveness of ICU follow-up clinics vs. standard-of-care in improving qualitative/clinical outcomes of ICU survivors and caregivers, with those receiving follow-up care hypothesized to have improved outcomes.

The intervention group will receive: 1) specialized follow-up care at 1- and 3-months following discharge, 2) information packages on expectations following discharge, and 3) diaries for the healthcare team, family, and patient to journal their experiences throughout recovery. The control group will receive generalized standard of care through their primary care provider. Focus groups will be used for qualitative assessment to elucidate what patients find most important for their recovery, using a patient-centred approach. Clinical assessments will evaluate neurocognitive function, quality of life, anxiety, depression, post-traumatic stress disorder, and resiliency among both ICU survivors and caregivers; chronic pain, fatigue, activities of daily living, lower extremity strength, polypharmacy, and hospital readmissions among ICU survivors; and caregiver burden and sleep quality among caregivers.

ICU survivorship extends beyond surviving the ICU. This program of research will unravel the aspects of follow-up care needed to mitigate the long-term impacts of PICS and improve patient and caregiver outcomes. This study is a first-step toward achieving this goal, by understanding barriers to successful recruitment, enrolment, data collection, and follow-up in this vulnerable cohort of ICU survivors and caregivers.

ELIGIBILITY:
Inclusion criteria - ICU survivors

1. Adult patients (age greater than or equal to 18 years)
2. Life expectancy greater than or equal to 6 months as determined by the attending physician
3. High risk for long-term functional sequelae following ICU discharge, defined as ICU stay greater than or equal to 4 days, or involving at least one of:

   * mechanical ventilation (any, i.e., invasive or non-invasive)
   * tracheostomy
   * delirium (defined as Confusion Assessment Method (CAM) positive or documented history of delirium in the patient's medical record by the clinical care team at some point during their ICU admission)
   * lack of access to a primary care physician for clinical follow-up
   * access to email or mail to complete follow-up questionnaires
   * presence of an informal caregiver

Inclusion criteria - Caregivers

1. Informal caregiver (e.g., spouse, offspring) for ICU survivor as defined above
2. Adult (age greater than or equal to 18 years)

Exclusion criteria - ICU survivors and caregivers

* Neurological or communication difficulties which would preclude completion of follow-up assessments or participation in focus groups
* Inability to speak or read English (required for completion of standardized questionnaires, clinical assessments, and for participation in focus groups)
* Failure to provide consent/failure to have consent provided by a substitute decision maker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Consent Rate | 6 months
  To determine the feasibility of a pragmatic RCT evaluating the impact of a post-ICU follow-up clinic intervention on clinical and qualitative patient and caregiver outcomes, as assessed via the following measure:
  Consent rate, measured as the proportion of eligible population who consent to participate
Feasibility - Enrolment Rate | 6 months
  To determine the feasibility of a pragmatic RCT evaluating the impact of a post-ICU follow-up clinic intervention on clinical and qualitative patient and caregiver outcomes, as assessed via the following measures:
  Enrolment rate, measured as the proportion of consented participants who are randomized
Feasibility - Follow-Up Rate | 6 months
  To determine the feasibility of a pragmatic RCT evaluating the impact of a post-ICU follow-up clinic intervention on clinical and qualitative patient and caregiver outcomes, as assessed via the following measures:
  Follow-up rate, measured as the proportion of enrolled participants who complete follow-up visits at 1-, 3-, and 6-months
Feasibility - Data Capture Rate | 6 months
  To determine the feasibility of a pragmatic RCT evaluating the impact of a post-ICU follow-up clinic intervention on clinical and qualitative patient and caregiver outcomes, as assessed via the following measures:
  Data capture rate, measured as the percentage of data elements acquired at each study time point
Feasibility - Rate of adverse events | 6 months
  To determine the feasibility of a pragmatic RCT evaluating the impact of a post-ICU follow-up clinic intervention on clinical and qualitative patient and caregiver outcomes, as assessed via the following measures:
  Rate of adverse events, assessed using the number of hospital and ICU readmissions, as well as the number of visits to the emergency department at 6 months.

SECONDARY OUTCOMES:
Qualitative impact of intervention | 6 months
  To determine the qualitative impact of a post-ICU follow-up care intervention on patients and caregivers, as assessed via qualitative analysis of focus group discussions.
Process evaluation | 6 months
  To perform a process evaluation of the multimodal ICU follow-up bundle of care intervention to understand the implementation, acceptability, content, barriers, and facilitators to use of diaries, informational materials, and the follow-up clinic.

OTHER OUTCOMES:
Neurocognition | 6 months
  Neurocognitive outcomes, as measured using the MoCA
Weight and BMI | 6 months
  To determine the effect of a post-ICU follow-up clinic intervention on changes in weight and body-mass index (BMI) following ICU discharge
Clinical Outcome | 6 months
  Frailty, as measured using the CFS
Quality of Life | 6 months
  Quality of life outcomes, as measured using the SF-36
Anxiety and mood | 6 months
  Anxiety and depression, as measured using the HADS
Post-traumatic stress | 6 months
  PTSD, as measured using the PTSS-14
Chronic pain | 6 months
  Chronic pain, as measured using the Chronic Pain Grade Scale (CPGS)
Fatigue | 6 months
  Chronic fatigue, as measured using the Fatigue Severity Scale (FSS)
Activities of daily living | 6 months
  Activities of daily living (ADLs), as measured using the Katz Index of ADLs
Instrumental activities of daily living | 6 months
  Instrumental ADLs, as measured using the Lawton IADL score
Physical function | 6 months
  Lower extremity strength, as measured using the 30-second Sit-to-Stand Test
Resiliency | 6 months
  Dyadic resiliency among ICU survivors and caregivers, as measured using the dyadic Connor-Davidson 10-item Resiliency Scale (CD-RISC-10)
Return to work | 6 months
  To determine the effect of a post-ICU follow-up clinic intervention on return to work by ICU survivors
Employment status of caregivers | 6 months
  Employment status relative to previous among caregivers

CONTACTS AND LOCATIONS:
Locations (1):
- Queen's University, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Jawa NA, Maslove DM, Sibley S, Muscedere J, Hunt M, Hanley M, Boyd T, Westphal R, Mathur S, Fakolade A, Tryon M, Boyd JG. IMPACT-ICU feasibility study: pragmatic mixed-methods randomised controlled trial of a follow-up care intervention for survivors of critical illness and caregivers. BMJ Open. 2025 Jan 2;15(1):e086799. doi: 10.1136/bmjopen-2024-086799. PMID 39753245